CLINICAL TRIAL: NCT06836180
Title: An Exploratory Study of Near-infrared Light Therapy for Mild to Moderate Alzheimer's Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024443
Record Dates: First submitted 2025-01-12; First posted 2025-02-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Once a day, once 30 minutes of near-infrared light treatment, 6 times a week for 96 weeks
  Interventions: Device: Near infrared light therapy

INTERVENTIONS:
Device: Near infrared light therapy — Once a day, once 30 minutes of near-infrared light treatment, 6 times a week for 96 weeks

SUMMARY:
This is an exploratory clinical study to evaluate the efficacy and safety of near-infrared light therapeutics in the treatment of mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
This experiment adopts a single-center, single-arm research design. All the patients who signed the informed consent were screened, and qualified subjects could only be enrolled to receive NIR therapy. This study plans to enroll 40 patients, all of whom meet the enrollment conditions will receive NIR therapy, and the treatment is arranged to be once a day, once a 30min NIR therapy, 6 times a week. The treatment lasted for 96 weeks, and follow-up and assessment were performed at baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks, 60 weeks, 72 weeks, 84 weeks, 96 weeks. During the first week of treatment, caregivers will be trained in the use of the NIR device, and after the training is complete, researchers will also provide remote guidance, making visits as needed. Changes in the 96-week ADAS-cog score from baseline were used as the primary endpoint to verify the efficacy and safety of the NIR device.

ELIGIBILITY:
Inclusion Criteria:

* 50 - 90 years old, no gender limitation;
* Meeting the National Institute on Aging and Alzheimer's Association (2011 NIA-AA) is likely the core clinical diagnostic criteria for Alzheimer's disease;
* The MMSE score is ≥ 12 and ≤ 26;
* The subjects should have primary school education or above and be able to complete the cognitive ability measurement and other tests stipulated in the protocol;
* If taking cognitive-improving medications, the dose must be stable for at least 12 weeks prior to enrollment (stable for at least 4 weeks with psychotropic medications);
* Participants themselves or their guardians voluntarily participate and sign the informed consent.

Exclusion Criteria:

* Any cognitive impairment or dementia not caused by Alzheimer's disease, or co-existing with a serious mental illness (schizophrenia, bipolar disorder, major depression, etc.);
* Currently taking anticoagulant drugs;
* A history of seizures or hemorrhagic stroke within 12 months;
* Allergic to sunlight or visible light or high sensitivity to head and neck skin;
* Severe head trauma or implants (bone nails, bone plates, excision, etc.);
* Malignant tumors;
* Any other medical condition that is not stabilized and adequately controlled (such as serious heart, respiratory, gastrointestinal, or kidney disease), or that the investigator believes may affect patient safety or interfere with the evaluation of the test;
* Persons addicted to alcohol or drugs;
* Women who are pregnant, nursing or planning a pregnancy;
* Participated in other clinical studies within 1 month before participating in this trial;
* Other conditions deemed unsuitable for clinical trial participation by the investigator.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's disease assessment scale-cognitive section(ADAS-Cog) | baseline, 96 weeks
  change from baseline on the Alzheimer's disease assessment scale-cognitive section(ADAS-Cog)

SECONDARY OUTCOMES:
ADAS-Cog | baseline,12 weeks,24 weeks,36 weeks,48 weeks, 60 weeks, 72 weeks, 84 weeks
  change from baseline on the Alzheimer's disease assessment scale-cognitive section(ADAS-Cog)
Mini Mental state Examination (MMSE) | baseline,12 weeks,24 weeks,36 weeks,48 weeks, 60 weeks, 72 weeks, 84 weeks, 96 weeks
  change from baseline on the Mini Mental state Examination (MMSE) score
Quantification of T-cell Subpopulation Proportions in Cerebrospinal Fluid (CSF) via Single-Cell RNA Sequencing | baseline, 12 weeks
  To determine the proportional abundance of T-cell subsets (e.g., CD4+, CD8+, regulatory T cells) within the cerebrospinal fluid (CSF) of patients using single-cell RNA sequencing (scRNA-seq).
Comprehensive Profiling of Glycolytic and Lipid Metabolic Substrates in Cerebrospinal Fluid (CSF) via Metabolomics | baseline, 12 weeks
  To quantify the concentrations of key metabolites involved in glycolysis (e.g., glucose, lactate, pyruvate) and lipid metabolism (e.g., free fatty acids, acylcarnitines, phospholipids) in cerebrospinal fluid (CSF) using liquid chromatography-tandem mass spectrometry (LC-MS/MS)-based metabolomics.
Quantification of Alzheimer's Disease (AD)-Associated Pathogenic Proteins in Cerebrospinal Fluid (CSF) via Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS) | baseline, 12 weeks
  To measure the concentration of AD-related neurotoxic proteins (e.g., amyloid-beta 42 [Aβ42], total tau, phosphorylated tau [p-tau181/217], neurofilament light chain [NfL]) in cerebrospinal fluid (CSF) using high-sensitivity liquid chromatography-tandem mass spectrometry (LC-MS/MS).

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China